CLINICAL TRIAL: NCT00735605
Title: Comparative Study Between Surgical and Non Surgical Treatment of Anismus in Patients With Symptoms of Obstructed Defecation
Brief Title: Comparative Study Between Surgical and Non Surgical Treatment of Anismus in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: ayman el nakeeb, mansour universty hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: anismus surgical and non
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obstructed Defecation; Anismus; Constipation
Keywords: obstructed defecation; constipation; puborectalis
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1:BFD (Active Comparator): The investigators used pressure based biofeedback training, using a perfused eight-channel polyvinyl catheter with a compliant balloon at the tip
  Interventions: Other: BFD
- 2 BTX A (Active Comparator): Injected with BTX-A in the left lateral position; anesthesia was not required
  Interventions: Other: BTX A
- 3: PDPR (Active Comparator): Inner half of puborectalis sling was divided on each side by using a scalpel NO
  Interventions: Procedure: PDPR

INTERVENTIONS:
Other: BFD — The investigators used pressure based biofeedback training, using a perfused eight-channel polyvinyl catheter with a compliant balloon at the tip
  Other Names: BIOFEEDBACK RETRAINING
  Arms: 1:BFD
Procedure: PDPR — A 2-3 cm curved incision is made on either side of the anal canal along its posterolateral aspect, each about 2.5 cm distance from the anal verge Fig(2). After that dissection in ischiorectal fossa was done till reaching the puborectalis sling from outside i.e. extrasphincteric approach . Using a right angle forceps the puborectalis sling is lifted up, guided by the contralateral index finger in the anal canal Fig(3). Nearly the inner half of puborectalis sling was divided on each side by using a scalpel NO. 11 Fig(4). Complete haemostasis was followed by skin closure without drain
  Other Names: PARTIAL DIVISION OF PUBORECTALIS
  Arms: 3: PDPR
Other: BTX A — A vial of Dysport, 500 u, (Dysport, Ipsen, United Kingdom) is dissolved in 2.5 ml isotonic saline Fig(1). A volume of 0.5 ml of dissolved toxin, i.e., 100 u Dysport, is injected in each patient
  Other Names: BOTILINUM TOXIN
  Arms: 2 BTX A

SUMMARY:
Comparative study between surgical and non surgical treatment of anismus in patients with symptoms of obstructed defecation.

Anismus is a significant cause of chronic constipation. This study came to compare the results of BFB training , BTX-A injection and PDPR in the treatment of anismus patients. Patients and methods: Seventy two anismus patients fulfilled Rome II criteria for functional constipation were included in this study. All patients underwent anorectal manometry, balloon expulsion test, defecography, and electromyography activity of the EAS. All patients had non relaxing puborectalis muscle.. The patients were randomized into three groups. Group I patients received biofeedback therapy, two times per week for about 1 month. Group II patients were injected with BTX- A. Group 111 partial division of puborectalis was done. Follow up was conducted weekly in the first month then monthly for about 1 year.

DETAILED DESCRIPTION:
Key words:

Obstructed defecation, chronic constipation, puborectalis, pelvic floor

ELIGIBILITY:
Inclusion Criteria:

* 60patients fulfilled Rome II criteria for functional constipation
* All patients were unresponsive to laxatives or enema use

Exclusion Criteria:

* Pregnant patients
* Patients with sphincteric defect
* Any patient proved to have colonic inertia by colon transit time
* Any patient with previous history of pelvic surgery e.g. mesh rectopexy
* Duhamel operation were excluded

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
improvement in bowel habit (regarding the straining severity, anorectal pain,number of weakly bowel movement,sensation of incomplete defecation and need of digitation or enema and using constipation score) | 1 year

SECONDARY OUTCOMES:
per rectal examination,manometeric relaxation,balloon expulsion,defecogram,EMG examination of anal sphincter to monitor any change in paradoxical contraction,recurrences,incontinence,complication | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: ayman elnakeeb, MD, Principal Investigator — MANSUORA UNIVERSITY HOSPITAL
Locations (1):
- Ayman Elnakeeb, Al Mansurah, Egypt

REFERENCES:
- [Background] Farid M, El Monem HA, Omar W, El Nakeeb A, Fikry A, Youssef T, Yousef M, Ghazy H, Fouda E, El Metwally T, Khafagy W, Ahmed S, El Awady S, Morshed M, El Lithy R. Comparative study between biofeedback retraining and botulinum neurotoxin in the treatment of anismus patients. Int J Colorectal Dis. 2009 Jan;24(1):115-20. doi: 10.1007/s00384-008-0567-0. Epub 2008 Aug 22. PMID 18719924
- [Result] Farid M, Youssef T, Mahdy T, Omar W, Moneim HA, El Nakeeb A, Youssef M. Comparative study between botulinum toxin injection and partial division of puborectalis for treating anismus. Int J Colorectal Dis. 2009 Mar;24(3):327-34. doi: 10.1007/s00384-008-0609-7. Epub 2008 Nov 29. PMID 19039596
- [Result] Maria G, Brisinda G, Bentivoglio AR, Cassetta E, Albanese A. Botulinum toxin in the treatment of outlet obstruction constipation caused by puborectalis syndrome. Dis Colon Rectum. 2000 Mar;43(3):376-80. doi: 10.1007/BF02258305. PMID 10733120
- [Result] Kamm MA, Hawley PR, Lennard-Jones JE. Lateral division of the puborectalis muscle in the management of severe constipation. Br J Surg. 1988 Jul;75(7):661-3. doi: 10.1002/bjs.1800750713. PMID 3416122
- [Result] Park UC, Choi SK, Piccirillo MF, Verzaro R, Wexner SD. Patterns of anismus and the relation to biofeedback therapy. Dis Colon Rectum. 1996 Jul;39(7):768-73. doi: 10.1007/BF02054442. PMID 8674369